CLINICAL TRIAL: NCT03311334
Title: A Phase 1b/2, Multicenter, Open-Label Study of DSP-7888 Dosing Emulsion in Combination With Immune Checkpoint Inhibitors Nivolumab or Pembrolizumab in Adult Patients With Advanced Solid Tumors
Brief Title: A Study of DSP-7888 Dosing Emulsion in Combination With Immune Checkpoint Inhibitors in Adult Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision to terminate development of the program.
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBI-DSP7888-102CI
Record Dates: First submitted 2017-10-09; First posted 2017-10-17 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-03

CONDITIONS: Renal Cell Carcinoma (RCC); Urothelial Carcinoma; Primary Peritoneal Cancer; Platinum-resistant Ovarian Cancer (PROC); Serous Epithelial Ovarian Cancer; Fallopian Tube Cancer
Keywords: DSP-7888; Nelatimotide; Adegramotide; immune checkpoint inhibitor; cancer vaccine; WT1; ICI; Wilms Tumor 1; Ombipepimut-S; nivolumab; Opdivo; pembrolizumab; Keytruda; Ovarian cancer; Platinum-resistant ovarian cancer; PROC; Serous epithelial ovarian cancer; High-grade serous epithelial ovarian cancer; HGSOC; Fallopian tube cancer; FTC; Peritoneal cancer; Primary peritoneal cancer; PPC; Renal cell carcinoma; Kidney cancer; RCC; Metastatic Renal Cell Carcinoma; Metastatic RCC; Metastatic kidney cancer; Advanced Renal Cell Carcinoma; Advanced RCC; Advanced kidney cancer; Urothelial carcinoma; Bladder cancer; Transitional cell carcinoma; UC; Metastatic urothelial carcinoma; Metastatic transitional cell carcinoma; Metastatic UC; Advanced urothelial carcinoma; Advanced UC; Advanced transitional cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma, Transitional Cell; Fallopian Tube Neoplasms; Wilms Tumor; Ovarian Neoplasms; Kidney Neoplasms; Urinary Bladder Neoplasms | interventions — Nivolumab; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DSP-7888 Dosing Emulsion in combination with Nivolumab (Experimental)
  Interventions: Drug: DSP-7888 Dosing Emulsion; Drug: Nivolumab
- DSP-7888 Dosing Emulsion in combination with Pembrolizumab (Experimental)
  Interventions: Drug: DSP-7888 Dosing Emulsion; Drug: Pembrolizumab

INTERVENTIONS:
Drug: DSP-7888 Dosing Emulsion — DSP-7888 Dosing Emulsion will be administered intradermally (ID) every 7 days until cycle 3, and then every 14 days for combination with Nivolumab arm or every 21 days for combination with Pembrolizumab arm.
  Other Names: Ombipepimut-S (adegramotide and nelatimotide)
Drug: Nivolumab — Nivolumab will be administered in the approved dose and schedule starting on Day 29 of the study.
  Other Names: Opdivo
  Arms: DSP-7888 Dosing Emulsion in combination with Nivolumab
Drug: Pembrolizumab — Pembrolizumab will be administered in the approved dose and schedule starting on Day 22 of the study.
  Other Names: Keytruda
  Arms: DSP-7888 Dosing Emulsion in combination with Pembrolizumab

SUMMARY:
This is a Phase 1b/2, open-label, multicenter study of DSP-7888 Dosing Emulsion in combination with checkpoint inhibitors (nivolumab or pembrolizumab) in adult patients with solid tumors, that consists of 2 parts: dose search part of the study (Phase 1b and Phase 1b Enrichment Cohort) and the dose expansion part of the study (Phase 2). In Phase 1b of this study there will be 2 arms: Arm 1 and Arm 2. In Arm 1, there will be 6 to 12 patients who will be dosed with DSP-7888 Dosing Emulsion and nivolumab and in Arm 2 there will be 6 to 12 patients who will be dosed with DSP-7888 Dosing Emulsion and pembrolizumab. In addition, an enrichment cohort of a further 10 patients who have locally advanced or metastatic Renal Cell Carcinoma or Urothelial Cancer with primary or acquired resistance to previous checkpoint inhibitors will be enrolled into Phase 1b of the study to help evaluate the preliminary antitumor activity of DSP-7888 Dosing Emulsion at the safe dose level identified in the dose-search part of the study, and will be dosed with DSP-7888 Dosing Emulsion and nivolumab, or DSP-7888 Dosing Emulsion and pembrolizumab, as per the investigator's preference. At the safe, recommended dose determined in Phase 1b, platinum-resistant ovarian cancer (PROC) patients will be enrolled in Phase 2 of the study with DSP-7888 Dosing Emulsion, exploring the combination with pembrolizumab (Arm 2). In Phase 2, approximately 40 patients with PROC will be initially enrolled; additional patients may be enrolled to further assess anti-tumor activities, but the total sample size will not exceed 60 patients. This brings the total maximum study population to approximately 84 patients.

ELIGIBILITY:
Inclusion Criteria Phase 1b:

Patients must fulfill each of the following requirements:

1. Phase 1b Dose Search Part Only: A histologically or cytologically confirmed cancer that is metastatic and is approved to be treated with nivolumab or pembrolizumab with the following origins:

   * Nivolumab: unresectable or metastatic melanoma, metastatic NSCLC, advanced RCC, recurrent or metastatic squamous cell carcinoma of the head and neck, locally advanced or metastatic urothelial carcinoma, hepatocellular carcinoma, MSI-H/dMMR colorectal cancer
   * Pembrolizumab: unresectable or metastatic melanoma, metastatic NSCLC, recurrent or metastatic squamous cell carcinoma of the head and neck, locally advanced or metastatic urothelial carcinoma, unresectable or metastatic MSI-H/dMMR solid tumors, recurrent locally advanced or metastatic gastric cancer or gastroesophageal junction adenocarcinoma, recurrent or metastatic cervical cancer

   In addition, the following requirements must be fulfilled:
   1. Patients must not be considered eligible for a potentially curative resection.
   2. Patients who are eligible for PD-1 therapy based on either criterion (i) or (ii) below:

   (i) Patients progressed on their prior treatment before initiating treatment on current study, OR (ii) Patients who are currently being treated with nivolumab or pembrolizumab and have achieved at least stable disease (SD), and who, in the judgment of their treating physicians, could benefit from the addition of DSP-7888 Dosing Emulsion vaccine to improve or maintain their response.

   Phase 1b Enrichment Cohort Only: Patients with locally advanced or metastatic RCC or urothelial carcinoma who have experienced disease progression per iRECIST (iCPD) during or within 3 months of last dose of the most recent prior anti-PD-1/ PD-L1-based treatment
2. Patients must be positive for at least 1 of the following human leukocyte antigens:

   1. HLA-A*02:01
   2. HLA-A*02:06
   3. HLA-A*24:02
   4. HLA-A*03:01
   5. HLA-B*15:01
3. ≥ 18 years of age
4. Eastern Cooperative Oncology group (ECOG) performance status of 0 or 1
5. Patients must be able to provide archival tumor tissue with sufficient tumor tissue, or patients must consent to undergo tumor biopsy to acquire sufficient tissue before first administration of study
6. Females of childbearing potential must have a negative serum pregnancy test
7. Male or female patients of child-producing potential must agree to use contraception or use prevention of pregnancy measures (true abstinence) during the study and for 6 months (for females and males alike) after the last dose
8. Total bilirubin of ≤ 2.0 mg/dL (≤ 3.0 mg/dL for patients with known Gilbert's syndrome)
9. Aspartate aminotransferase (AST) ≤ 3.0 × the upper limit of normal (ULN) or < 5 × ULN if considered to be due to liver metastases
10. Alanine transaminase (ALT) ≤ 3.0 × the upper limit of normal (ULN) or < 5 × ULN if considered to be due to liver metastases
11. Glomerular Filtration Rate > 40 mL/min
12. Multigated acquisition (MUGA) scan or echocardiogram with left ventricular ejection fraction (LVEF) > 40%
13. Life expectancy ≥ 3 months
14. Patients must be willing to provide a signed and dated ICF

Exclusion Criteria Phase 1b:

Patients with any of the following will be excluded from the study:

1. Anticancer chemotherapy (including molecular targeted drugs), immunotherapy, radiotherapy, or investigational agents within 4 weeks of the first dose of DSP 7888 Dosing Emulsion
2. Major surgery within 4 weeks prior to study treatment
3. Patients who have received a live vaccine within 4 weeks prior to the first dose
4. Any known, untreated brain metastases; patients with treated brain metastases must be clinically stable for 4 weeks after completion of treatment for brain metastases and have radiographic image documentation of stability. Patients must have no clinical symptoms from brain metastases and not have required systemic corticosteroids > 10 mg/day prednisone or equivalent for at least 2 weeks prior to the first dose of study drug
5. Patients who have multifocal glioblastoma
6. Pregnant or breastfeeding
7. Patients who have an active autoimmune disease requiring immunosuppression > 10 mg/day prednisone or equivalent a. Patients with controlled hyperthyroidism must be negative for thyroglobulin and thyroid peroxidase antibodies and thyroid stimulating immunoglobulin prior to study drug administration
8. Patients who have interstitial lung disease or active, non-infectious pneumonitis
9. Known hypersensitivity to a component of protocol therapy:

   1. Patients with known hypersensitivity to any of the components of DSP-7888 Dosing Emulsion.
   2. Patients with known hypersensitivity to nivolumab or pembrolizumab are excluded from receiving combination therapy that includes the agent to which they are hypersensitive
10. Uncontrolled concurrent illness including, but not limited to: ongoing or active, uncontrolled bacterial, viral, or fungal infections requiring systemic therapy; clinically significant non-healing or healing wounds; symptomatic congestive heart failure; unstable angina pectoris; severe and/or uncontrolled cardiac arrhythmia; significant pulmonary disease; or, psychiatric illness/social situations that would limit compliance with study requirements
11. Patients with a history of another primary cancer with the exception of: (a) curatively resected non-melanoma skin cancer; (b) curatively treated cervical carcinoma in situ; (c) localized prostate cancer not requiring systemic therapy; and d) any another cancer from which the patient has been disease free for ≥ 2 years that, in the opinion of the Investigator and medical monitor for the Sponsor, will not affect patient outcome in the setting of the current diagnosis
12. Patients who have a QTcF (QT corrected based on Fridericia's equation) interval > 480 msec (CTCAE = Grade 2) or other factors that increase the risk of QT prolongation or arrhythmic events (e.g. heart failure, hypokalemia, family history of long QT interval syndrome) at screening
13. Patients who have a medical history of frequent or sustained ventricular ectopy
14. Patients who have, in the opinion of the treating Investigator, any concurrent conditions that could pose an undue medical hazard or interfere with the interpretation of the study results
15. Known history of human immunodeficiency virus (HIV) infection, active hepatitis B, or untreated hepatitis C
16. Patients who have baseline signs and symptoms consistent with clinically significant, decreased pulmonary function: (1) blood saturation oxygen level (SpO2) < 90% at rest on room air; (2) dyspnea at rest or required supplemental oxygen within 2 weeks of study enrollment

Inclusion Criteria Phase 2:

Patients eligible for inclusion must meet all of the following criteria:

1. Patients must be female ≥ 18 years of age, able to understand study procedures, and subsequently agreed to participate in the study by providing a written informed consent obtained prior to any prescreening and screening procedures that are not standard of care 2.

Patients must be positive for at least 1 of the following human leukocyte antigens (HLA):

a. HLA-A*02:01 b. HLA-A*02:06 c. HLA-A*24:02 d. HLA-A*03:01 e. HLA-B*15:01

3. Patients must have histologically diagnosed ovarian, fallopian tube, or primary peritoneal cancer with predominantly high-grade (Grade 2 or 3) serous epithelial features 4. Patients must be considered platinum resistant to last administered platinum-based therapy, defined as patient relapsed within 6 months after last dose of platinum-based therapy 5. Patients must have completed at least 1 but no more than 4 prior lines of therapy for serous epithelial ovarian, fallopian tube, or primary peritoneal cancer;

1. Maintenance is not considered a separate line of treatment (even if patients with BRCA mutation positive received PARP-inhibitor following induction therapy with a platinum doublet including bevacizumab, etc.)
2. Neoadjuvant and adjuvant systemic therapy will be counted as one line of therapy
3. Patients must have received at least one platinum-based therapy

   6. Patients must have progression disease after last therapy and have measurable disease according to RECIST (v1.1).

   7. Patients must have an ECOG performance status of 0 or 1. 8. Patients must have adequate organ function, defined as follows:

Hematological:

1. Absolute neutrophil count (ANC) ≥ 1,500/μL (without granulocyte-colony stimulating factor (G-CSF))
2. Platelets ≥ 100,000/μL (without transfusion)
3. Hemoglobin ≥ 9.0 g/dL (without transfusion)

Renal:

a. Serum Creatinine OR estimated glomerular filtration rate using the Cockcroft-Gault equation ≤ 1.5 × the upper limit of normal (ULN) OR 40 mL/min using the Cockcroft-Gault equation for patients with creatinine levels > 1.5 × ULN

Hepatic:

1. Serum total bilirubin ≤ 1.5 ULN
2. Aspartate aminotransferase (AST) and alanine transaminase (ALT) ≤ 2.5 × ULN OR ≤ 5 × ULN for patients with liver metastases

Cardiac:

1. Multigated acquisition (MUGA) scan or echocardiogram with left ventricular ejection fraction (LVEF) ≥ 40%.
2. QTcF (QT corrected based on Fridericia's equation) interval < 480 msec

Coagulation:

1. International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 × ULN
2. Activated Partial Thromboplastin Time (aPTT) or Partial Thromboplastin Time (PTT) ≤ 1.5 × ULN

   9. Patients must provide a fresh tissue biopsy, if medically feasible, or archival tissue as either a formalin-fixed and paraffin embedded FFPE) block or newly sectioned tissue on charged slides (equivalent to approximately 8-23 slides sectioned at 4-5μm thickness) 10. Patients of childbearing potential must have a negative serum or urine pregnancy test at screening 11. Patients must be either postmenopausal, free from menses > 12 months, surgically sterilized, or willing to use adequate contraception to prevent pregnancy or must agree to abstain from heterosexual activity throughout the study, starting with enrollment through 6 months after the last dose of study treatment 12. Life expectancy ≥ 3 months 13. Patients who had stayed on the last treatment for at least 12 weeks without any evidence of progression

Exclusion Criteria Phase 2:

Patients with any of the following will be excluded from the study:

1. Primary platinum refractory patients defined as patients who experienced disease progression during the treatment with first-line platinum therapy
2. Patients with a known, untreated brain metastasis. Patients with treated brain metastases must be clinically stable for 4 weeks after completion of treatment for brain metastases and have radiographic image documentation of stability. Patients must have no clinical symptoms from brain metastases and not have required systemic corticosteroids > 10 mg/day prednisone or equivalent for at least 4 weeks prior to the first dose
3. Patients who have received prior treatment with any other anti-PD-1, or PD-L1 or PD-L2 agent or an antibody or a small molecule targeting other immuno-regulatory receptors or mechanisms (examples of such drugs include but are not limited to antibodies against CTLA-4, LAG-3, IDO, PD-L1, IL-2R, GITR)
4. Patients who have received prior treatment with any other Wilms Tumor 1 (WT1)-related agents including peptide vaccine, dendric cell vaccine, and gene therapy
5. Patients who have received treatment for ovarian cancer within the following time frame prior to the first dose of the study

   1. Cytotoxic chemotherapy, hormonal therapy; ≤ 3 weeks
   2. Targeted therapy except for monoclonal antibody; ≤ 3 weeks
   3. Immune therapy, biologic therapy (e.g. antibodies); ≤ 4 weeks
   4. Other investigational agents: ≤ 4 weeks
   5. Radiation therapy (except for localized radiotherapy for analgesic purpose) ≤ 4 weeks
   6. Radiation therapy (localized radiotherapy for analgesic purpose) ≤ 1 week
   7. Major surgery regardless of reason ≤ 4 weeks.
6. Patients who have received a live vaccine within 4 weeks prior to the first dose.
7. Any known additional malignancy that is progressing or requires active treatment with the exception of:

   1. curatively treated basal cell or squamous cell carcinoma of skin
   2. curatively treated superficial bladder cancer, carcinoma in situ of the cervix,
   3. any another cancer from which the patient has been disease free for ≥ 3 years without any active treatment that, in the opinion of the Investigator and medical monitor for the Sponsor, will not affect patient's outcome in the setting of the current diagnosis.
8. Patients who have not recovered to < CTCAE Grade 2 or baseline from toxic effect (with exception of alopecia and/or neuropathy) of prior cancer therapy.
9. Patients who have an active autoimmune disease requiring systemic immunosuppression in excess of physiologic maintenance dose of corticosteroids (> 10 mg/day prednisone or equivalent) or any other forms of immunosuppressive therapy within 7 days prior to the first dose of study drug.
10. Positive serology for HIV infection, active hepatitis B, or hepatitis C
11. Patients who have a known history of bacillus tuberculosis (TB).
12. Patients with impaired cardiac function or clinically significant cardiac disease;

    * New York Hospital Association Class III or IV cardiac disease, including preexisting clinically significant ventricular arrythmia, congestive heart failure, or cardiomyopathy
    * Unstable angina pectoris ≤ 6 months before study participation
    * Myocardial infarction or stroke ≤ 6 months before study participation
13. Patients who have an interstitial lung disease or a history of pneumonitis that required oral or intravenous glucocorticoids to assist with management
14. Patients with active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
15. Patients with any psychiatric condition, substance abuse disorder, or social situation that would interfere with a patient's cooperation with the study requirements and schedule
16. Patients with any condition that would, in the investigator's judgment, interfere with full participation including administration of study drugs, attending required visits or interfere with interpretation of study data
17. Patients who are pregnant or breastfeeding
18. Patients who have known hypersensitivity to DSP-7888 Dosing Emulsion, pembrolizumab, their components, or their excipients
19. Patient has dyspnea at rest (CTCAE ≥ Grade 3) or has required supplemental oxygen within 2 weeks of study enrollment
20. Patients with history of bowel obstruction related to underlying disease within 3 months prior to the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-11-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (17):
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UC San Francisco Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - AdventHealth Cancer Institute, Orlando, Florida
  - Decatur Memorial Hospital, Decatur, Illinois
  - Horizon Oncology Research, Lafayette, Indiana
  - Norton Cancer Institute, Louisville, Kentucky
  - St Vincent Frontier Cancer Center, Billings, Montana
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - UC Health, LLC, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - West Cancer Clinic, Germantown, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Summit Cancer Centers, Spokane, Washington
- Canada (2):
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - SMBD Jewish General Hospital, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who died, withdrew consent to survival follow up or were lost to follow up were considered to have completed the study.
Groups:
- Phase 1b - DSP-7888 10.5 mg + Nivolumab 240 mg: DSP-7888 Dosing Emulsion 10.5mg administered intradermally (ID) every 7 days until cycle 3, and then every 14 days for combination with Nivolumab 240mg IV.
- Phase 1b - DSP-7888 10.5 mg + Pembrolizumab 200 mg/8mL; Phase 2 - DSP-7888 10.5mg + Pembrolizumab 200mg/8mL: DSP-7888 Dosing Emulsion 10.5mg administered intradermally (ID) every 7 days until cycle 3, and then every 21 days for combination with Pembrolizumab 200mg/8mL IV starting on cycle 1 day 22 every 3 weeks.
Period: Overall Study
Arm/Group | Phase 1b - DSP-7888 10.5 mg + Nivolumab 240 mg | Phase 1b - DSP-7888 10.5 mg + Pembrolizumab 200 mg/8mL | Phase 2 - DSP-7888 10.5mg + Pembrolizumab 200mg/8mL
Started | 7 | 9 | 31
Completed | 7 | 9 | 31
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1b - Arm 1: DSP-7888 Dosing Emulsion in combination with Nivolumab
  DSP-7888 Dosing Emulsion: DSP-7888 Dosing Emulsion will be administered intradermally (ID) every 7 days until cycle 3, and then every 14 days for combination with Nivolumab arm or every 21 days for combination with Pembrolizumab arm.
  Nivolumab: Nivolumab will be administered in the approved dose and schedule starting on Day 29 of the study.
- Phase 1b - Arm 2: DSP-7888 Dosing Emulsion in combination with Pembrolizumab
  DSP-7888 Dosing Emulsion: DSP-7888 Dosing Emulsion will be administered intradermally (ID) every 7 days until cycle 3, and then every 14 days for combination with Nivolumab arm or every 21 days for combination with Pembrolizumab arm.
  Pembrolizumab: Pembrolizumab will be administered in the approved dose and schedule starting on Day 22 of the study.
- Phase 2 - Ombipepimut-S + Pembrolizumab: The Phase 2 dose of ombipepimut-S Dosing Emulsion will be the recommended dose as determined in the Phase 1b Arm 2 part of the study.
- Total: Total of all reporting groups
Arm/Group | Phase 1b - Arm 1 | Phase 1b - Arm 2 | Phase 2 - Ombipepimut-S + Pembrolizumab | Total
Number analyzed (Participants) | 7 | 9 | 31 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 13 | 22
  >=65 years | 3 | 4 | 18 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 31 | 37
  Male | 5 | 5 | 0 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 7 | 8 | 27 | 42
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 9 | 31 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events and Serious Adverse Events
Time Frame: From the date of signing informed consent until 30 days after last dose for an average of 3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b - Arm 1 | Phase 1b - Arm 2 | Phase 2 - Ombipepimut-S + Pembrolizumab
Number analyzed (Participants) | 7 | 9 | 31
Participants | 7 | 9 | 31

2. Primary Outcome: Determination of the Recommended Phase 2 Dose (RP2D) by Assessing Dose-limiting Toxicities (DLTs).
Description: The RP2D was based on the data collected during phase 1b.
Time Frame: 28 days
Population: Only data from arm 2 of phase 1b were analyzed to determine the RP2D.
Measure: Number; unit: mg
Arm/Group | Phase 1b - Arm 2
Number analyzed (Participants) | 9
mg | 10.5

3. Primary Outcome: Phase II: The Objective Response Rate (ORR) of DSP-7888 Dosing Emulsion Administered With Pembrolizumab in Patients With Platinum-resistant Ovarian Cancer (PROC).
Description: Defined as the proportion of patients who have achieved confirmed Complete Response or Partial Response by RECIST v1.1 based on investigator assessment.
Time Frame: Radiographic imaging every 6 weeks for 24 weeks and then every 12 weeks until progression for an average of 12 months
Population: Sponsor's decision to terminate the study, hence data for determination of ORR were not collected.
Arm/Group | Phase 2 - Ombipepimut-S + Pembrolizumab
Number analyzed (Participants) | 0

4. Secondary Outcome: Phase Ib: The Objective Response Rate (ORR) of DSP-7888 Dosing Emulsion Administered With Pembrolizumab or Nivolumab
Description: Defined as the proportion of patients who have achieved confirmed complete response (CR) or partial response (PR) evaluated using RECIST v1.1 and iRECIST.
Time Frame: At 4 weeks for the nivolumab arm and at 6 weeks for the pembrolizumab arm and then at Weeks 12, 18, and 24 after the first dose of the DSP-7888 dosing emulsion
Population: Sponsor's decision to terminate study. No data were collected and analyzed.
Arm/Group | Phase 1b - Arm 1 | Phase 1b - Arm 2
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Phase Ib: The Disease Control Rate (DCR) of DSP-7888 Dosing Emulsion Administered With Pembrolizumab or Nivolumab
Description: Defined as the percentage of patients who have achieved best overall response (BOR) of complete response (CR), partial response (PR), or stable disease (SD) per RECIST v1.1 and iRECIST.
Time Frame: as for outcome 4
Population: Sponsor's decision to terminate study. No data were collected and analyzed.
Arm/Group | Phase 1b - Arm 1 | Phase 1b - Arm 2
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Phase Ib: Assessment of the Duration of Response (DOR) of Ombipepimut-S in Combination With Nivolumab or Pembrolizumab
Description: DOR is defined as the time from first documentation of response until the time of first documentation of disease progression by RECIST v1.1 and iRECIST or death by any cause.
Time Frame: At week 4 for patients on the nivolumab arm and week 6 for patients on the pembrolizumab arm. Thereafter weeks 12, 18 and 24 and every 12 weeks until progression or death.
Population: Sponsor's decision to terminate study. Therefore no data were collected nor analyzed.
Arm/Group | Phase 1b - Arm 1 | Phase 1b - Arm 2
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Phase Ib: Progression-free Survival (PFS) of DSP-7888 Dosing Emulsion Administered With Pembrolizumab or Nivolumab
Description: The percentage of participants with a complete response or partial response who have measurable disease at baseline imaging.
Time Frame: Radiographic imaging every 6 weeks for 24 weeks and then every 12 weeks until progression for an average of 12 months
Population: Sponsor's decision to terminate study. No data were collected and analyzed.
Arm/Group | Phase 1b - Arm 1 | Phase 1b - Arm 2
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Phase Ib: The 6-month Progression-free Survival (PFS) Rate of Ombipepimut-S in Combination With Nivolumab or Pembrolizumab
Description: Defined as the proportion of patients who neither progressed by RECIST (v.1.1) nor died before 6 months (24 weeks) from the first study treatment
Time Frame: 6 months
Population: Sponsor's decision to terminate study. No data were collected or analyzed.
Arm/Group | Phase 1b - Arm 1 | Phase 1b - Arm 2
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Phase Ib: Percentage of Patients With Overall Survival (OS) When Treated With Ombipepimut-S in Combination With Nivolumab or Pembrolizumab
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1b - Arm 1 | Phase 1b - Arm 2
Number analyzed (Participants) | 7 | 9
percentage of participants | 0 | 0

10. Secondary Outcome: Phase II: Assessment of the Duration of Response (DOR) of Ombipepimut-S in Combination With Pembrolizumab
Description: Defined as the time from the first documentation of a response (CR or PR) until time of first documentation of disease progression by RECIST v1.1 or death by any cause.
Time Frame: Radiographic imaging every 6 weeks for 24 weeks and then every 12 weeks until progression up to 24 months.
Population: Sponsor's decision to terminate the study. Hence data were not collected nor analyzed.
Arm/Group | Phase 2 - Ombipepimut-S + Pembrolizumab
Number analyzed (Participants) | 0

11. Secondary Outcome: Phase II: Disease Control Rate of Ombipepimut-S in Combination With Pembrolizumab
Description: Defined as the percentage of patients who have achieved best overall response (BOR) of complete response, partial response, or stable disease per RECIST (v.1.1)
Time Frame: Radiographic imaging every 6 weeks for 24 weeks and then every 12 weeks until progression, up to 24 months.
Population: Sponsor's decision to terminate the study. Hence data were not collected nor analyzed.
Arm/Group | Phase 2 - Ombipepimut-S + Pembrolizumab
Number analyzed (Participants) | 0

12. Secondary Outcome: Phase II: Assessment of the Progression-free Survival (PFS) of Ombipepimut-S in Combination With Pembrolizumab
Description: Defined as the time from the date of the first dose of study treatment to the earlier date of assessment of progression by RECIST v.1.1, or death by any cause
Time Frame: Radiographic imaging every 6 weeks for 24 weeks and then every 12 weeks until progression, up to 24 months
Population: Sponsor's decision to terminate the study. Hence data were not collected nor analyzed.
Arm/Group | Phase 2 - Ombipepimut-S + Pembrolizumab
Number analyzed (Participants) | 0

13. Secondary Outcome: Phase II: 6-month Progression-free Survival (PFS) of Ombipepimut-S in Combination With Pembrolizumab
Description: PFS is defined as the time from the date of the first dose of study treatment to the earlier date of assessment of progression by RECIST (v.1.1), or death by any cause
Time Frame: 6 months
Population: Sponsor's decision to terminate the study. Hence data were not collected nor analyzed.
Arm/Group | Phase 2 - Ombipepimut-S + Pembrolizumab
Number analyzed (Participants) | 0

14. Secondary Outcome: Phase II: Overall Survival of Patients Treated With Ombipepimut-S in Combination With Pembrolizumab
Description: Defined as the time from the date of first dose of study treatment to the date of death by any cause
Time Frame: Every 3 months from last dose of study treatment up to 24 months.
Population: Sponsor's decision to terminate the study. Hence data were not collected nor analyzed.
Arm/Group | Phase 2 - Ombipepimut-S + Pembrolizumab
Number analyzed (Participants) | 0

15. Secondary Outcome: Phase II: Immune Objective Response Rate (iORR) of Ombipepimut-S in Combination With Pembrolizumab
Description: Defined as the percentage of patients who have achieved confirmed immune complete response (iCR) or immune partial response (iPR), evaluated using iRECIST based on investigator's assessment.
Time Frame: Up to 24 months
Population: Sponsor's decision to terminate the study. Hence data were not collected nor analyzed.
Arm/Group | Phase 2 - Ombipepimut-S + Pembrolizumab
Number analyzed (Participants) | 0

16. Secondary Outcome: Phase II: Immune Disease Control Rate (iDCR) of Ombipepimut-S in Combination With Pembrolizumab
Description: Defined as the percentage of patients who have achieved best overall response of iCR, iPR, or immune stable disease (iSD), per iRECIST
Time Frame: Up to 24 months
Population: Sponsor's decision to terminate the study. Hence data were not collected nor analyzed.
Arm/Group | Phase 2 - Ombipepimut-S + Pembrolizumab
Number analyzed (Participants) | 0

17. Secondary Outcome: Phase II: Immune Progression-free Survival (iPFS) of Ombipepimut-S in Combination With Pembrolizumab
Description: Defined as the time from the date of the first dose of study treatment to the earlier date of assessment of progression by iRECIST or death by any cause
Time Frame: Up to 24 months
Population: Sponsor's decision to terminate the study. Hence data were not collected nor analyzed.
Arm/Group | Phase 2 - Ombipepimut-S + Pembrolizumab
Number analyzed (Participants) | 0

18. Secondary Outcome: Phase II: Immune Duration of Response (iDOR) of Ombipepimut-S in Combination With Pembrolizumab
Description: Defined as the time from the first documentation of response (iCR or iPR) until time of first documentation of disease progression by iRECIST, or death by any cause
Time Frame: Up to 24 months
Population: Sponsor's decision to terminate the study. Hence data were not collected nor analyzed.
Arm/Group | Phase 2 - Ombipepimut-S + Pembrolizumab
Number analyzed (Participants) | 0

19. Secondary Outcome: Phase II: Evaluation of the Safety and Tolerability of Ombipepimut-S in Combination With Pembrolizumab
Description: Demonstrated by the number of participants with adverse events and serious adverse events
Time Frame: Up to 24 months
Population: Sponsor's decision to terminate the study. Hence data were not collected nor analyzed.
Arm/Group | Phase 2 - Ombipepimut-S + Pembrolizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Serious and Other Adverse Events were assessed from the date of first treatment through 30 days of the last administration of study drug, an average of 12 months. All-Cause Mortality was assessed from the date of first treatment until death, an average of 24 months.
Arm/Group | Phase 1b - Arm 1 | Phase 1b - Arm 2 | Phase 2 - Ombipepimut-S + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 1/7 | 0/9 | 1/31
Serious Adverse Events (participants affected / at risk) | 3/7 | 5/9 | 8/31
Other Adverse Events (participants affected / at risk) | 7/7 | 9/9 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b - Arm 1 (N=7) | Phase 1b - Arm 2 (N=9) | Phase 2 - Ombipepimut-S + Pembrolizumab (N=31)
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Spinal Cord Compression (Nervous system disorders) | 1 | 0 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Urine Output Decreased (Investigations) | 0 | 1 | 1
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Pnemonia (Infections and infestations) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pericardial Effusion (Cardiac disorders) | 1 | 1 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1 | 1
Cardiac Tamponade (Cardiac disorders) | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0
Large Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 2
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 5
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b - Arm 1 (N=7) | Phase 1b - Arm 2 (N=9) | Phase 2 - Ombipepimut-S + Pembrolizumab (N=31)
Constipation (Gastrointestinal disorders) | 2 | 3 | 7
Nausea (Gastrointestinal disorders) | 1 | 2 | 13
Pyrexia (Gastrointestinal disorders) | 0 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1 | 8
Dental Caries (Gastrointestinal disorders) | 1 | 0 | 0
Diabetic Ketoacidosis (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 7
Ascites (Gastrointestinal disorders) | 0 | 0 | 5
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 5
Flatulence (Gastrointestinal disorders) | 0 | 0 | 3
Ileus (Gastrointestinal disorders) | 0 | 0 | 2
Large Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 2
Early Satiety (Gastrointestinal disorders) | 0 | 1 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 3
Oral Pain (Gastrointestinal disorders) | 1 | 1 | 1
Injection Site Reaction (General disorders) | 7 | 9 | 23
Decreased Appetite (General disorders) | 2 | 5 | 4
Fatigue (General disorders) | 2 | 4 | 15
Localised Oedema (General disorders) | 0 | 0 | 2
Pain in Extremity (General disorders) | 1 | 2 | 2
Dysphonia (General disorders) | 1 | 1 | 0
Hypophosphataemia (General disorders) | 2 | 0 | 1
Abdominal Pain Upper (General disorders) | 0 | 0 | 3
Chest Discomfort (General disorders) | 1 | 0 | 1
Infusion Related Reaction (General disorders) | 1 | 0 | 0
Night Sweats (General disorders) | 0 | 1 | 0
Non-cardiac Chest Pain (General disorders) | 0 | 1 | 2
Periorbital Oedema (General disorders) | 1 | 0 | 0
Peripheral Swelling (General disorders) | 0 | 1 | 0
Sunburn (General disorders) | 0 | 1 | 0
Tooth Infection (General disorders) | 1 | 0 | 0
Abdominal Pain (General disorders) | 0 | 0 | 10
Abdominal Distension (General disorders) | 0 | 0 | 7
Dry Mouth (General disorders) | 0 | 0 | 3
Injection Site Pain (General disorders) | 7 | 9 | 23
Oedema peripheral (General disorders) | 2 | 1 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Injection Site Pain (General disorders) | 0 | 0 | 3
Pain (General disorders) | 0 | 0 | 3
Headache (Nervous system disorders) | 2 | 1 | 9
Insomnia (Nervous system disorders) | 1 | 2 | 3
Dizziness (Nervous system disorders) | 0 | 2 | 2
Paraesthesia (Nervous system disorders) | 2 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 2
Hot Flush (Nervous system disorders) | 1 | 0 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Pyrexia (Nervous system disorders) | 0 | 0 | 7
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 5
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Amylase Increased (Investigations) | 1 | 0 | 0
Blood Urine (Investigations) | 1 | 0 | 0
Fibrin D Dimer Increased (Investigations) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 3 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Blood Creatinine Increased (Investigations) | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Platelet Count Decreased (Investigations) | 0 | 1 | 0
Vitamin B12 Deficiency (Investigations) | 0 | 1 | 0
Weight Increased (Investigations) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 3
Lymphocyte Count Decreased (Investigations) | 0 | 0 | 3
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 2
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 2
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 2
Gamma-glutamyltransferase Increased (Investigations) | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Weight Decreased (Investigations) | 0 | 2 | 4
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 7
Conjunctival Haemorrhage (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Chest Pain (Cardiac disorders) | 2 | 0 | 0
Electrocardiogram QT Prolonged (Cardiac disorders) | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4
Abdominal Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 5
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 2
Influenza Like Illness (Infections and infestations) | 1 | 1 | 5
Sinusitis (Infections and infestations) | 2 | 0 | 0
Herpes Zoster (Infections and infestations) | 1 | 0 | 0
Nail Disorder (Infections and infestations) | 1 | 0 | 0
Nail Infection (Infections and infestations) | 1 | 0 | 0
Otitis Media (Infections and infestations) | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 4
Corona Virus Infection (Infections and infestations) | 0 | 0 | 2
Oral Infection (Infections and infestations) | 1 | 0 | 0
Myringitis (Infections and infestations) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 2 | 2
Confusional State (Psychiatric disorders) | 0 | 2 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Psychomotor Hyperactivity (Psychiatric disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 2 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 2 | 0
Arthropod Bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fibula Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal Cord Compression (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 2
Hypersensitivity (Injury, poisoning and procedural complications) | 2 | 0 | 1
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 1 | 1
Dry Eye (Eye disorders) | 0 | 1 | 0
Eye Pain (Eye disorders) | 0 | 1 | 0
Photopsia (Eye disorders) | 0 | 1 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT03311334/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT03311334/SAP_001.pdf